CLINICAL TRIAL: NCT03930901
Title: Impact of Health Education Learning Package Against Intestinal Parasitic Infections Among Orang Asli Schoolchildren in Malaysia
Brief Title: Impact of Health Education Learning Package Against Intestinal Parasitic Infections Among Orang Asli Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Nabil Ahmed Mohammed Nasr, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202016000190-85
Record Dates: First submitted 2019-04-05; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Intestinal Parasitic Infections; Knowledge, Attitudes, Practice
Keywords: Intestinal Parasitic Infections; Soil-transmitted helminth infections; Health education
MeSH Terms: conditions — Behavior; Health Education

STUDY DESIGN:
Intervention Model Description: Two groups; intervention group that involved schools where HELP will be administered and control group that involved schools that will not receive health education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Children in this group were examined for intestinal parasites and then treated accordingly. Then, health education learning package (HELP) was introduced to children in the selected schools. The package involved different items and activities during the study period, e.g. comic booklet on the intestinal parasitic infections, stand banners, posters, lectures, songs, drawing competition, puppet show, lectures, with a toolkit that involved soap, slipper (plastic clogs shoes), & nail clipper).
  Interventions: Other: Health education learning package
- Control (No Intervention): Children in this group were examined for intestinal parasites and then treated accordingly. They were follow up for 6 months.

INTERVENTIONS:
Other: Health education learning package — Health education learning package (HELP) was introduced to children in the selected schools. The package involved different items and activities during the study period, e.g. comic booklet on the intestinal parasitic infections, stand banners, posters, lectures, songs, drawing competition, puppet show, lectures, with a toolkit that involved soap, slipper (plastic clogs shoes), & nail clipper).
  Other Names: HELP
  Arms: Intervention

SUMMARY:
A health education learning package (HELP) has been improved and evaluated for its impact against intestinal parasitic infections among Orang Asli schoolchildren in West Malaysia. 13 schools were allocated into two groups (intervention and control groups) and the impact of HELP was evaluated after 3 and 6 months of baseline assessment and HELP intervention.

DETAILED DESCRIPTION:
This study was conducted to evaluate the impact of an improved health education learning package (HELP) against intestinal parasitic infections among Orang Asli schoolchildren in West Malaysia. The package has been tested by a pilot study in 2013 among children in 2 schools in Pahang state.

In the current study, HELP package has been improved and children from 13 primary schools in 11 districts of six states in Peninsular Malaysia were allocated into two groups (intervention and control groups) and the impact of HELP was evaluated after 3 and 6 months of baseline assessment and HELP intervention.

The evaluation involved soil-transmitted helminth infections and intestinal protozoa infections.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2 - 6
* Orang Asli ethnicity
* Schools exclusively for Orang Asli

Exclusion Criteria:

* Grade 1
* Chronic sever diseases
* no consent
* schools for mixed population groups

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1142 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Re-infection rate of intestinal parasitic infections using multiple parasitological and molecular diagnostic techniques | 6 months
  Prevalence rate of Intestinal parasitic infections before and after health education

SECONDARY OUTCOMES:
Intensity rate of intestinal parasitic infections using multiple parasitological and molecular diagnostic techniques | 6 months
  Intensity rate of Intestinal parasitic infections before and after health education

CONTACTS AND LOCATIONS:
Overall Officials: Hesham M Al-Mekhlafi, PhD, Study Director — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Delaimy AK, Al-Mekhlafi HM, Lim YA, Nasr NA, Sady H, Atroosh WM, Mahmud R. Developing and evaluating health education learning package (HELP) to control soil-transmitted helminth infections among Orang Asli children in Malaysia. Parasit Vectors. 2014 Sep 2;7:416. doi: 10.1186/1756-3305-7-416. PMID 25179100